CLINICAL TRIAL: NCT01521143
Title: A Randomized Trial of Cvac (Autologous Dendritic Cells Pulsed With Recombinant Human Fusion Protein [Mucin 1-glutathione S-transferase] Coupled to Oxidized Polymannose) as Maintenance Treatment in Patients With Epithelial Ovarian Cancer (EOC) in Complete Remission Following First-line Chemotherapy (A) and Patients With EOC in Second Remission (B)
Brief Title: Cvac as Maintenance Treatment in Patients With Epithelial Ovarian Cancer in Complete Remission Following First-line Chemotherapy or Second-line Treatment
Acronym: CANVAS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to company restructuring and changes in drug development priorities.
Sponsor: Prima BioMed Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAN-004
Record Dates: First submitted 2012-01-17; First posted 2012-01-30 (Estimated); Results first posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Epithelial Ovarian Cancer
Keywords: EOC
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — CCV-AV protocol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Part A - Cvac (Experimental): Participants received intradermal injections of Cvac given at 4-week intervals for the first 3 doses, and then every 12 weeks for 3 additional doses, for a total of 6 doses over 44 weeks. Each injection had an approximate concentration of 60 × 10^6 viable dendritic cells/mL.
  Interventions: Biological: Cvac
- Part A - Placebo (Placebo Comparator): Participants received intradermal injections of placebo given at 4-week intervals for the first 3 doses, and then every 12 weeks for 3 additional doses, for a total of 6 doses over 44 weeks.
  Interventions: Biological: Placebo
- Part B - Cvac (Experimental): Participants received intradermal injections of Cvac given at 4-week intervals for the first 3 doses, and then every 12 weeks for 3 additional doses, for a total of 6 doses over 44 weeks. Each injection had an approximate concentration of 60 × 10^6 viable dendritic cells/mL.
  Interventions: Biological: Cvac
- Part B - Observational standard of care (No Intervention): Participants in this group did not receive any treatment during the study.

INTERVENTIONS:
Biological: Cvac — Injections were done at 4 anatomical sites, 1 injection in each of the upper portions of both arms and both thighs.
  Arms: Part A - Cvac; Part B - Cvac
Biological: Placebo — Injections were done at 4 anatomical sites, 1 injection in each of the upper portions of both arms and both thighs.
  Placebo consisted of the Cvac formulation buffer (5% HSA, 10% DMSO) with 0.9% simethicone provided in 1 mL vials that had been cryopreserved and stored at the manufacturing facility.
  Arms: Part A - Placebo

SUMMARY:
As < 10% of the necessary patients required by the protocol were recruited and the data were not intended to support a labeling claim, it was determined that the abbreviated clinical study report (CSR) was the appropriate reporting format. No efficacy analyses were performed as the trial was terminated early with incomplete enrollment of < 10%.

The purpose of this study is to determine if an investigational cell therapy called Cvac can help epithelial ovarian cancer (EOC) from returning when administered to patients who are in complete remission after surgical removal of their tumor followed by standard first-line (Part A) or second-line (Part B) chemotherapy. Following remission, patients will undergo leukapheresis for the manufacture of the study agent. After completion of chemotherapy and confirmation of remission, patients will enter the treatment phase of the study.

DETAILED DESCRIPTION:
This study proposes a nontoxic immunotherapeutic approach to extend overall survival in patients in complete remission. Most patients with ovarian cancer achieve complete clinical remission after optimal debulking surgery and first-line platinum-based chemotherapy. However, most patients, despite high response rates to first-line treatment, will relapse and undergo subsequent chemotherapy. Generally, the progression-free interval between treatments becomes shorter with each relapse, and the patient eventually dies of the disease.

For production of Cvac, each patient's cells were enriched using cell separation techniques. The patient's cells were cultured for 5 days with granulocyte-macrophage colony-stimulating factor (GM-CSF) and interleukin-4 (IL-4) in AIM V® serum-free tissue culture medium (Thermo Fisher Scientific) to cultivate the growth of dendritic cells (DC). The culture was pulsed overnight with the antigen (mannosylated mucin 1 fusion protein [M-FP]) to arm the DCs to the specific mucin 1 antigen. After harvesting, the M-FP-pulsed DCs were formulated as a finished product (Cvac) in 1 mL aliquots, diluted in 5% human serum albumin (HSA) and 10% dimethyl sulfoxide (DMSO) at an approximate concentration of 60 × 10^6 viable DCs/mL. The vials were cryopreserved and stored in the vapor phase of liquid nitrogen at the manufacturing facility.

Different participants were enrolled in the 2 parts of the study.

Part A

To be eligible for participation, patients were diagnosed with stage III or IV epithelial ovarian cancer, underwent optimal debulking surgery (≤ 1 cm of residual disease), underwent platinum and taxane chemotherapy, with or without bevacizumab, and had a tumor that overexpressed mucin 1, as well as met all other study inclusion and exclusion criteria at screening.

Patients who met all study inclusion and exclusion criteria were randomized in a 1:1 double-blinded fashion to either the Cvac (active) group or the placebo (control) group. After randomization, patients underwent mononuclear cell (MNC) collection for production of the study agent and then began first-line chemotherapy. After completion of chemotherapy and confirmation of complete clinical and radiological remission (Baseline), patients were entered into the treatment phase of the study.

A total of 76 patients were recruited and randomized at centers in Europe, North America, and Australia.

Part B

To be eligible for participation, patients had first-line platinum-based chemotherapy with a complete response lasting for at least 6 months prior to relapse and achieved second remission following standard platinum-based second-line chemotherapy with or without a second bulk-reducing surgery, and had a tumor that over-expressed mucin 1, as well as met all other study inclusion and exclusion criteria.

Patients who met all study inclusion and exclusion criteria were randomized in a 1:1 fashion to either the Cvac (active) group or the observational standard of care (control) group. After randomization, only patients randomized to Cvac underwent MNC collection for production of the study agent. After confirmation of no evidence of disease at the Baseline visit, patients were entered into the treatment phase of the study.

A total of 15 patients were recruited and randomized at centers in Europe.

ELIGIBILITY:
Part A: First Remission

Inclusion Criteria (Part A):

1. Females ≥ 18 years of age at screening with a confirmed diagnosis of Stage III or IV epithelial ovarian, primary peritoneal, or fallopian tube cancer.
2. Undergone optimal debulking surgery, defined as ≤ 1 cm of residual tumor.
3. Undergone standard platinum and taxane first-line chemotherapy.
4. Signed an informed consent form (ICF).
5. Completed study procedures within the study timelines.
6. Mucin 1-positive tumor as determined by central immunohistopathology.
7. Adequate renal function in the opinion of the investigator based on serum creatinine and/or glomerular filtration rate.
8. Adequate liver function, defined as serum glutamic oxaloacetic transaminase/aspartate aminotransferase (SGOT/AST) and serum glutamic pyruvic transaminase/alanine aminotransferase (SGPT/ALT) ≤ 2× ULN and serum bilirubin ≤ 1.5 × ULN, unless Gilbert's syndrome had been previously confirmed for the patient.
9. Adequate bone marrow function, defined as white blood cells (WBCs) ≥ 3.0 K/µL, absolute neutrophil count (ANC) ≥ 1.5 × 109/L, hemoglobin ≥ 9 g/dL, and platelets ≥ 100 × 109/L.
10. Life expectancy of at least 12 months at the time of screening as judged by the investigator.
11. Not pregnant, and if of childbearing potential, agreed to use a highly effective method of birth control (implanted, injectable, or oral combination hormonal method alone or in possible combinations, intrauterine device, vasectomized partner, or abstinence) prior to study entry, for the duration of the study, and for 3 months after the last dose of study agent. Male partners of a study patient must use a condom in addition to the acceptable method of contraception for the female partner, as specified above.

Exclusion Criteria (Part A):

1. Non-epithelial ovarian cancer, including ovarian germ cell, sarcoma, mixed Müllerian tumors, or mucinous carcinoma of the peritoneum.
2. Malignancy other than epithelial ovarian cancer, except those that had been in complete response for a minimum of 3 years, and except carcinoma in-situ of the cervix or basal cell and squamous cell carcinomas of the skin that had been adequately treated.
3. Treatment with any investigational product (for any condition) within 4 weeks of screening.
4. Concurrent systemic treatment with steroids or other immunosuppressant agents at a dose considered by the investigator to be higher than a standard physiological dose.
5. Evidence of severe or uncontrolled cardiac disease, including myocardial infarction or unstable angina within 6 months of screening, congestive heart failure, or ventricular arrhythmias requiring medication.
6. Clinically significant abnormalities as measured by electrocardiogram (ECG).
7. Active uncontrolled infection.
8. Uncontrolled hypertension.
9. Diagnosed immunodeficiency or autoimmune disorder.
10. Infection with human immunodeficiency virus (HIV) or hepatitis C virus (HCV), or active and infectious hepatitis B virus (HBV) infection.
11. Pregnant or lactating.
12. Evidence or history of central nervous system metastasis.
13. Known hypersensitivity to any of the components of the study agent.
14. Active or latent infection with Mycobacterium tuberculosis in any body tissue (especially renal and/or lung).
15. Any other health condition that would preclude participation in the study in the judgment of the principal investigator.

Part B: Second Remission

Inclusion Criteria (Part B):

1. Females ≥ 18 years of age at screening with a confirmed diagnosis of epithelial ovarian, fallopian tube, or peritoneal cancer.
2. Underwent standard cytoreductive surgery and first-line chemotherapy containing platinum before first relapse and were in complete remission for at least 6 months prior to relapse.
3. Relapsed once and then underwent standard platinum-based second-line chemotherapy (at least 3 cycles is required) with or without a second bulk-reducing surgery.
4. Second remission defined as:

   1. No definitive evidence of disease (NED) on computed tomography (CT) or magnetic resonance imaging (MRI) of the abdomen and pelvis;
   2. CA-125 ≤ upper limit of normal (ULN) or 90% reduction in CA-125 since start of second-line chemotherapy;
   3. Negative physical exam (ie, no clinical signs).
5. Life expectancy ≥ 3 months in the opinion of the investigator.
6. Signed an informed consent form (ICF).
7. Willing and able to complete study procedures within the expected study timelines.
8. Mucin 1-positive tumor as determined by central immunohistopathology.
9. Histologically documented EOC, fallopian tube, or peritoneal cancer (patients with pseudomyxoma, mesothelioma, unknown primary tumor, sarcoma, or neuroendocrine histology, with borderline ovarian cancer, ie, patients with low malignant potential tumors, and with clear cell or mucinous histology are excluded).
10. Adequate end-organ and hematological function as defined by:

    1. Adequate bone marrow function: white blood cells (WBCs) ≥ 3.0 K/µL, absolute neutrophil count (ANC) ≥ 1.5 × 109/L, hemoglobin ≥ 9 g/dL, and platelets ≥ 100 × 109/L.
    2. Adequate renal function, defined as serum creatinine ≤ 1.5 × ULN.
    3. Adequate liver function, defined as serum glutamic oxaloacetic transaminase/aspartate aminotransferase (SGOT/AST) and serum glutamic pyruvic transaminase/alanine aminotransferase (SGPT/ALT) ≤ 2 × ULN and serum bilirubin ≤ 1.5 × ULN.
11. Generally well-controlled blood pressure with systolic blood pressure ≤ 140 mmHg and diastolic blood pressure ≤ 90 mmHg prior to randomization (antihypertensive medications are permitted). Low-dose chronic hormonal or steroidal treatments are also permitted.
12. Not pregnant, and if of childbearing potential, agrees to use a highly effective method of birth control (implanted, injectable, or oral combination hormonal method alone or in possible combinations, intrauterine device, vasectomized partner, or abstinence) prior to study entry, for the duration of the study, and for 3 months after the last dose of study agent. Male partners of a study patient must use a condom in addition to the acceptable method of contraception for the female partner, as specified above.
13. Eastern Cooperative Oncology Group (ECOG) status of 0 or 1 (applicable at the baseline visit only).

Exclusion Criteria (Part B):

1. More than 2 previous lines of chemotherapy for EOC, fallopian tube, or peritoneal cancer.
2. Primary platinum-refractory or platinum-resistant disease (ie, patients who progress prior to cessation of induction therapy [platinum refractory] or recur within 6 months after cessation [platinum resistant]).
3. Treatment with any investigational product (for any condition) within 4 weeks of screening. Enrolled in or has not completed at least 28 days of treatment (prior to screening) since ending another investigational device or drug treatment, or currently receiving other investigational treatments.
4. Concurrent systemic treatment with steroids or other immunosuppressant agents at a dose considered by the investigator to be higher than a standard physiological dose.
5. Evidence of severe or uncontrolled cardiac disease, including myocardial infarction or unstable angina within 6 months of screening, congestive heart failure, or ventricular arrhythmias requiring medication.
6. Diagnosed immunodeficiency or autoimmune disorder.
7. Infection with human immunodeficiency virus (HIV) or hepatitis C virus (HCV), or active and infectious hepatitis B virus (HBV) infection.
8. Pregnant or lactating.
9. Evidence or history of central nervous system metastasis.
10. Known hypersensitivity to any of the components of the study agent.
11. Any unresolved persistent toxicities from prior systemic therapy that are either Grade 3 or Grade 4 (except alopecia) per the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
12. Intent to treat patient with both an anti-angiogenesis therapy (such as bevacizumab) and a poly (ADP-ribose) polymerase (PARP) inhibitor as part of maintenance therapy. Only one or the other are permitted while the patient is on study and must be started between the Baseline visit and Visit 1 (first treatment visit) if it will be used as part of the patient's maintenance therapy regimen.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2012-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - LAC-USC Medical Center, Los Angeles, California
  - Collaborative Research Group, Boynton Beach, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - University Gynecologic Oncology, Atlanta, Georgia
  - Women's Cancer Center, Morristown, New Jersey
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Australia (2):
  - Greenslopes Private Hospital, Greenslopes
  - Royal Brisbane and Women's Hospital, Herston

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Different participants were enrolled in the 2 parts of the study.
Period: Overall Study
Arm/Group | Part A - Cvac | Part A - Placebo | Part B - Cvac | Part B - Observational Standard of Care
Started | 40 | 36 | 8 | 7
Received Treatment | 20 | 20 | 3 | 4
Completed | 11 | 10 | 0 | 0
Not Completed | 29 | 26 | 8 | 7

BASELINE CHARACTERISTICS:
Population: Part A - Safety population: All randomized participants who received at least 1 dose of Cvac or placebo.
  Part B - Safety population: All randomized participants who received at least 1 dose of Cvac (Cvac group) or were evaluated at least once (observational standard of care group).
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A - Cvac | Part A - Placebo | Part B - Cvac | Part B - Observational Standard of Care | Total
Number analyzed (Participants) | 20 | 20 | 3 | 4 | 47
Age, Customized [Number; unit: Participants]
  45-65 years of age | 20 | 20 | 3 | 4 | 47
Gender [Count of Participants; unit: Participants]
  Female | 20 | 20 | 3 | 4 | 47
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A - Overall Survival
Description: Overall survival was defined as the number of days from Baseline to the date of death from any cause.
Time Frame: Baseline to the end of the study (up to 3 years, 2 months)
Population: Intent-to-treat population: All participants who were randomized to a treatment group. The data for this Outcome Measure were not analyzed since the study was terminated early.
Arm/Group | Part A - Cvac | Part A - Placebo | Part B - Cvac | Part B - Observational Standard of Care
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Part A - Time to Next Treatment
Description: Time to next treatment was defined as the number of days from Baseline to the date when the next treatment for epithelial ovarian cancer was started.
Time Frame: Baseline to the end of the study (up to 3 years, 2 months)
Population: as for outcome 1
Arm/Group | Part A - Cvac | Part A - Placebo | Part B - Cvac | Part B - Observational Standard of Care
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Part A - Progression-free Survival
Description: Progression-free survival was defined as the number of days from Baseline and the documented disease progression as defined by response evaluation criteria in solid tumors (RECIST) or death, whichever occurred earlier. Disease progression was defined as any measurable new lesion(s) that were accurately measured in at least 1 dimension. Any new lesion(s) with a minimum size of 20 mm were deemed as unequivocal (ie, clear or definite) progression. Any new lesion(s) with a minimum size of 15 mm but smaller than 20 mm were considered equivocal progression and had to be confirmed by a follow-up radiological procedure.
Time Frame: Baseline to the end of the study (up to 3 years, 2 months)
Population: as for outcome 1
Arm/Group | Part A - Cvac | Part A - Placebo | Part B - Cvac | Part B - Observational Standard of Care
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Part B - Overall Survival
Description: Overall survival was defined as the number of days from Baseline to the date of death from any cause.
Time Frame: Baseline to the end of the study (up to 3 years, 2 months)
Population: as for outcome 1
Arm/Group | Part A - Cvac | Part A - Placebo | Part B - Cvac | Part B - Observational Standard of Care
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Part B - Time to Next Treatment
Description: as for outcome 2
Time Frame: Baseline to the end of the study (up to 3 years, 2 months)
Population: as for outcome 1
Arm/Group | Part A - Cvac | Part A - Placebo | Part B - Cvac | Part B - Observational Standard of Care
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Part B - Progression-free Survival
Description: as for outcome 3
Time Frame: Baseline to the end of the study (up to 3 years, 2 months)
Population: as for outcome 1
Arm/Group | Part A - Cvac | Part A - Placebo | Part B - Cvac | Part B - Observational Standard of Care
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: Part A - Safety population: All randomized participants who received at least 1 dose of Cvac or placebo.
  Part B - Safety population: All randomized participants who received at least 1 dose of Cvac (Cvac group) or were evaluated at least once (observational standard of care group).
Arm/Group | Part A - Cvac | Part A - Placebo | Part B - Cvac | Part B - Observational Standard of Care
Serious Adverse Events (participants affected / at risk) | 5/20 | 7/20 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 17/20 | 13/20 | 2/3 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - Cvac (N=20) | Part A - Placebo (N=20) | Part B - Cvac (N=3) | Part B - Observational Standard of Care (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fat necrosis (General disorders) | 1 | 0 | 0 | 0
Hernia (General disorders) | 1 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 0
Herpes dermatitis (Infections and infestations) | 1 | 0 | 0 | 0
Poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Biopsy liver (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Stoma care (Surgical and medical procedures) | 1 | 0 | 0 | 0
Lymphocele (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - Cvac (N=20) | Part A - Placebo (N=20) | Part B - Cvac (N=3) | Part B - Observational Standard of Care (N=4)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 1 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0
Abdomianl pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lip blister (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 4 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0
Chills (General disorders) | 2 | 1 | 0 | 0
Edema (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 0 | 0
Feeling hot (General disorders) | 0 | 1 | 0 | 0
Hernia (General disorders) | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 2 | 0 | 1 | 0
Infusion site erythema (General disorders) | 0 | 1 | 0 | 0
Infusion site pain (General disorders) | 0 | 1 | 0 | 0
Injection site discomfort (General disorders) | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 5 | 4 | 0 | 0
Injection site hematoma (General disorders) | 1 | 0 | 0 | 0
Injection site nodule (General disorders) | 2 | 2 | 0 | 0
Injection site pain (General disorders) | 3 | 2 | 0 | 0
Injection site reaction (General disorders) | 2 | 2 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 1 | 0
Local swelling (General disorders) | 0 | 1 | 0 | 0
Nodule (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For study centers in Australia, no publication of the study results may be made until publication of the results of the study from all centers or until 2 years after study completion, whichever is sooner. For study centers in the USA, no submission for publication or public disclosure of the results by will be made until the results from all centers have been received and analyzed by the sponsor, or the multi-center study has been terminated or abandoned at all centers.